CLINICAL TRIAL: NCT01695928
Title: Effect of Low-energy Extracorporeal Shock Waves on Orthodontic Tooth Movement and Miniscrew Stability
Brief Title: Effect of Shock Waves on Tooth Movement and Miniscrew Stability
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Frank Falkensammer, DMD,DMS, DMD,DMS, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESWT2
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Mesial Movement of Teeth; Miniscrew Stability
Keywords: Velocity; Location; Periodontal status
MeSH Terms: conditions — Mesial Movement of Teeth | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extracorporeal shockwave therapy (ESWT) (Active Comparator): Active treatment
  Interventions: Device: Extracorporeal shockwave therapy
- ESWT Placebo (Placebo Comparator): No extracoporeal shockwave therapy
  Interventions: Device: ESWT placebo

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — 1000 impulses
  Other Names: Orthogold 100 MTS
  Arms: Extracorporeal shockwave therapy (ESWT)
Device: ESWT placebo — 0 impulses, acoustic effect
  Other Names: Orthogold 100 MTS
  Arms: ESWT Placebo

SUMMARY:
The low-energy extracorporal shockwave is a scientifically approved method to activate respectively increase bone-turnover processes especially in orthopedic medicine. The aim of this clinical study is to apply this effect in orthodontic dentistry and evaluate the orthodontic tooth movement respectively miniscrew stability clinically.

This randomized clinical study is carried out in orthodontic patients undergoing space closure therapy at the university clinic of dentistry. During this period the tooth movement rate as well as the miniscrew stability are evaluated consecutively chairside.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients which don´t fulfill the exclusion criteria

Exclusion Criteria:

* disease (syndroms,infections,...) which influence the bone turnover and the oral health
* medication, which influences the bone turnover and the oral health
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Orthodontic tooth movement | 4 months

SECONDARY OUTCOMES:
Miniscrew stability | 4 months

OTHER OUTCOMES:
Periodontal status | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans P Bantleon, Prof, M.D., Study Chair — Bernhard Gottlieb University Clinic of Dentistry, Department of Orthodontics
Locations (1):
- Bernhard Gottlieb University clinic of Dentistry, Vienna, Vienna, Austria

REFERENCES:
- [Result] Sathishkumar S, Meka A, Dawson D, House N, Schaden W, Novak MJ, Ebersole JL, Kesavalu L. Extracorporeal shock wave therapy induces alveolar bone regeneration. J Dent Res. 2008 Jul;87(7):687-91. doi: 10.1177/154405910808700703. PMID 18573992
- [Result] Martini L, Giavaresi G, Fini M, Torricelli P, de Pretto M, Schaden W, Giardino R. Effect of extracorporeal shock wave therapy on osteoblastlike cells. Clin Orthop Relat Res. 2003 Aug;(413):269-80. doi: 10.1097/01.blo.0000073344.50837.cd. PMID 12897619
- [Result] Hazan-Molina H, Kaufman H, Reznick ZA, Aizenbud D. [Orthodontic tooth movement under extracorporeal shock wave therapy: the characteristics of the inflammatory reaction--a preliminary study]. Refuat Hapeh Vehashinayim (1993). 2011 Jul;28(3):55-60, 71. Hebrew. PMID 21939106
- [Derived] Falkensammer F, Rausch-Fan X, Arnhart C, Krall C, Schaden W, Freudenthaler J. Impact of extracorporeal shock-wave therapy on the stability of temporary anchorage devices in adults: a single-center, randomized, placebo-controlled clinical trial. Am J Orthod Dentofacial Orthop. 2014 Oct;146(4):413-22. doi: 10.1016/j.ajodo.2014.06.008. PMID 25263143